CLINICAL TRIAL: NCT06664008
Title: The Effect of Probiotic and Zinc Supplementation in Patients With Gastroesophageal Reflux Disease
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Christina Medhat, Assistant Lecturer, British University In Egypt
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: FMASUR200/2024
Record Dates: First submitted 2024-10-27; First posted 2024-10-29 (Actual); Last update posted 2024-10-29 (Actual); Status verified 2024-10

CONDITIONS: Gastro-oesophageal Reflux Disease
MeSH Terms: conditions — Gastroesophageal Reflux | interventions — Proton Pump Inhibitors; Probiotics; Zinc

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Group 1: PPI alone (Active Comparator): Proton pump inhibitor
  Interventions: Drug: PPI (proton pump inhibitor)
- Group 2 (PPI+Probiotic) (Experimental): Proton pump inhibitor and Probiotic
  Interventions: Drug: PPI (proton pump inhibitor); Drug: Probiotic
- Group 3: PPI+Zinc (Experimental): Proton pump inhibitor and Zinc
  Interventions: Drug: PPI (proton pump inhibitor); Drug: Zinc
- Group 4: PPI+Probiotic and Zinc (Experimental): Proton pump inhibitor, Zinc and Probiotic
  Interventions: Drug: PPI (proton pump inhibitor); Drug: Probiotic; Drug: Zinc

INTERVENTIONS:
Drug: PPI (proton pump inhibitor) — It reduces stomach acid production and manage GERD symptoms
Drug: Probiotic — Live microorganisms, primarily bacteria and yeast, that are believed to provide health benefits when consumed in adequate.
  Arms: Group 2 (PPI+Probiotic); Group 4: PPI+Probiotic and Zinc
Drug: Zinc — Zinc used a supplement due to its role in decreasing inflammation of the gastroesophageal reflux disease.
  Arms: Group 3: PPI+Zinc; Group 4: PPI+Probiotic and Zinc

SUMMARY:
Introduction:

Gastroesophageal reflux disease (GERD) is a common digestive disorder affecting the esophagus and gastro-duodenum, presenting symptoms such as acid reflux and heartburn. GERD's incidence, symptoms, and prognosis are heavily influenced by diet and lifestyle factors. Current management of GERD involves lifestyle modifications (e.g., weight loss, dietary changes) and pharmacologic agents like proton pump inhibitors (PPIs), histamine-2-receptor blockers (H2 B), antacids, and medications that affect gastrointestinal motility (Kröner et al., 2021).

Background on Probiotics and Zinc:

Probiotics are non-pathogenic microorganisms that, when administered in adequate amounts, offer several health benefits, including improvement in conditions associated with inflammation and gut health. Probiotics, often of the Lactobacillusand Bifidobacterium species, interact with gut microbiota, enhance barrier function, and modulate immune responses (Cheng & Ouwehand, 2020; Kröner et al., 2021). Probiotics have been linked to reduced levels of inflammatory mediators, such as cytokines, and are recognized for their anti-inflammatory and antioxidant properties (Sharifi-Rad et al., 2020; Wang et al., 2017).

Zinc, specifically Zinc L-carnosine, exhibits antioxidant, cytokine modulation, and membrane-stabilizing properties, acting as a mucosal cytoprotective and anti-inflammatory agent (Efthymakis & Neri, 2022). Previous studies suggest that the combination of probiotics and zinc may be beneficial for gut health, but there is limited data on their effects on GERD symptoms, inflammation, and oxidative stress.

Study Aim:

To evaluate the effect of probiotics and zinc on GERD symptoms and to explore their potential antioxidant and anti-inflammatory effects.

Patients and Methods:

Study Design:

This is a prospective controlled randomized comparative study conducted at El-Demerdash Hospital, Ain Shams University Hospitals.

Ethical Considerations:

The study has received ethical approval from the Research Ethics Committee of the Faculty of Pharmacy, Ain Shams University, and the Scientific Research Ethics Committee at the Faculty of Medicine, Ain Shams University. It adheres to the Declaration of Helsinki and is registered on ClinicalTrials.gov.

Participants:

Inclusion Criteria: Adults aged 18-74 years with esophagitis confirmed by gastroscopy and GERD symptoms.

Exclusion Criteria: Allergy to study medications, pregnancy, severe renal or liver insufficiency, history of myocardial infarction, stroke, malignant tumors, and certain gastrointestinal conditions or surgeries.

Sample Size Calculation:

The study is designed to detect a large effect size (f = 0.4) for zinc and probiotic effects using G*Power software. A total of 120 patients will be recruited (30 per group) to account for a 15% dropout rate.

Study Groups:

Group I (Control): PPI (Omeprazole 40 mg daily). Group II: PPI + probiotic. Group III: PPI + zinc. Group IV: PPI + probiotic and zinc.

Methodology:

Participants will undergo baseline assessments, including medical history, gastroscopy, and measurement of gastrointestinal hormones, inflammatory markers (IL-6, IL-12, CRP), and oxidative stress markers (MDA). The same assessments will be repeated at the study's end after 4 weeks. Follow-up assessments will occur biweekly, and patients will be contacted between visits to monitor side effects.

Outcomes:

Primary Outcome: Change in Gastrointestinal Symptom Rating Scale (GSRS) scores and gastrin hormone levels before and after treatment.

Secondary Outcomes:

Anti-inflammatory effect (IL-6, IL-12, CRP levels). Antioxidant effect (MDA levels).

Statistical Analysis:

Data will be analyzed using SPSS. Statistical significance is set at p ≤ 0.05. Continuous variables will be expressed as mean ± SD or median (interquartile range), depending on distribution, and analyzed using appropriate tests (e.g., T-test or Mann-Whitney U test).

This study aims to provide insights into the potential benefits of probiotics and zinc in managing GERD symptoms and their anti-inflammatory and antioxidant effects, filling a current gap in the literature.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18-74 years; (both male and female).
* Esophagitis that might be confirmed by gastroscopy.
* Patients with confirmed symptoms of GERD N.B.: The typical clinical presentation of GERD is heartburn and regurgitation. Heartburn is defined as a retrosternal burning sensation or discomfort that may radiate into the neck and typically occurs after the ingestion of meals or when in a reclined position. Regurgitation is a retrograde migration of acidic gastric contents into the mouth or hypopharynx . GERD can also present with various other symptoms that include dysphagia, odynophagia, belching, epigastric pain, and nausea.

Exclusion Criteria:

* Allergy or potential allergy to the study medications.
* Pregnancy.
* Patients with CrCl< 20 ml/min or on dialysis.
* Patients with myocardial infarction, stroke, or malignant tumour.
* Patients with liver insufficiency (liver enzymes > 2*upper limit of normal)
* Heart Failure or ECG (electrocardiogram) abnormalities
* Gastroscopy that revealed any of the following diseases within the last 2 months: bleeding, esophageal and gastric varices, upper gastrointestinal malignant lesions.
* A history of gastroesophageal or duodenal surgery.

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-11-01 (Estimated); Primary Completion 2025-03-01 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
Change in Gastrointestinal Symptom Rating Scale (GSRS) | 1 month
  •The primary efficacy variable will be the change in Gastrointestinal Symptom Rating Scale (GSRS) score before and after treatment (reflecting the patient's experience of the dyspepsia symptoms during the preceding weeks: pain, heartburn, acid reflux, hunger, pain, nausea, stomach rumbles, stomach swelling, belching, bloating, constipation, diarrhea, and interchange between constipation and diarrhea) as well as the effect on gastrin hormone level.

SECONDARY OUTCOMES:
Anti-inflammatory effect will be measured through the markers (Interleukin-6 (IL-6), Interleukin-12 (IL-12) and CRP levels. | 1 month
Antioxidant effect measured through oxidative stress marker as (MAD). | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Nagwa A Sabri, Study Director — Ain Shams University

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR